CLINICAL TRIAL: NCT00653432
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of a Single Injection Cross-Linked Sodium Hyaluronate to Provide Symptomatic Relief of Osteoarthritis of the Knee
Brief Title: Safety and Effectiveness of Monovisc® Injection for Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Monovisc-0702
Record Dates: First submitted 2008-03-05; First posted 2008-04-07 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis
Keywords: Monovisc®; Hyaluronic Acid Gel; Injection; Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monovisc® (Experimental): Injectable Hyaluronic Acid Gel
  Interventions: Device: Monovisc®
- Saline (Placebo Comparator): 0.9% Sterile Saline
  Interventions: Other: Saline

INTERVENTIONS:
Device: Monovisc® — Intra-articular injection
  Other Names: Sodium Hyaluronate; Hyaluronic Acid Gel
  Arms: Monovisc®
Other: Saline — 0.9% Sterile Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether intra-articular injection of Monovisc® hyaluronic acid provides symptomatic relief of osteoarthritis of the knee.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo controlled prospective study will assess the safety and effectiveness of a single intra-articular injection of Monovisc® in providing symptomatic relief of pain caused by idiopathic osteoarthritis (OA) of the knee as compared to a placebo comparator injection of sterile saline.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or Female
* Age 35 to 75 years
* Body Mass Index (BMI) 20 to 40 kg/m2
* Willing and able to provide informed consent
* Willing to limit analgesic use to acetaminophen 7 days prior to and 12 weeks after injection
* Not pregnant or lactating
* Previous conservative treatment regimen for osteoarthritis (OA)
* Diagnosis of idiopathic OA of the index knee
* OA symptoms for >= 6 months
* Index knee Kellgren-Lawrence (K-L) grade of II or III
* Index knee Baseline Summed WOMAC Pain Score >= 200mm and < 400mm after NSAID washout
* Contralateral Knee K-L grade 0, I or II
* Contralateral Knee Baseline WOMAC Pain Score < 150mm after NSAID washout

Main Exclusion Criteria:

* Joint disorders which could interfere with treatment effectiveness
* Joint disorders which could interfere with study assessments
* Arthroscopy of either knee within 3 months of screening
* Open surgery of index knee within 12 months of screening
* Open surgery of contralateral knee within 3 months of screening
* Injection of Hyaluronic Acid (HA) in either knee within 6 months of screening
* Injection of steroid in index knee within 3 months of screening
* Any pre-treatment contraindication for injection or aspiration of the index knee, including cutaneous infection, intra-articular infection, knee deformity or condition which may jeopardize sterility or delivery of injection
* Synovial fluid aspirate volume > 20 milliliters (mL)
* Visual appearance of synovial fluid that contraindicates injection
* Index knee range of motion < 90 degrees
* Subject participation in other research study within 30 days of screening
* Subject unwilling to maintain active lifestyle, exercise program and body weight similar to that during 3 months prior to screening for duration of study
* Unwilling to maintain constant dosage of oral glucosamine or chondroitin sulfate for duration of study, if applicable
* Other medication or treatments that could interfere with study injection or assessments
* Allergy to gram positive bacterial products or intolerance of acetaminophen
* Active fibromyalgia
* Peripheral neuropathy severe enough to interfere with evaluation of either knee
* Vascular insufficiency severe enough to interfere with evaluation of the subject
* Hemiparesis involving either lower extremity
* Systemic bleeding disorder
* Other conditions which may adversely affect the success of the procedure

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schmitz, MD, Study Director — Prometrika, LLC
Locations (31):
- United States (30):
  - Clinical Research Consultants, Hoover, Alabama
  - Novara Clinical Research, Mesa, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Tuscon Orthopaedic Institute, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Summit Clinical Research, Aurora, Colorado
  - Boulder Medical Center, Boulder, Colorado
  - Colorado Orthopedic Consultants, Englewood, Colorado
  - Plancher Orthopaedic and Sports Medicine, Cos Cob, Connecticut
  - Community Research Foundation, Miami, Florida
  - Tampa Medical Clinic, Tampa, Florida
  - Resurgens Orthopedics, Cumming, Georgia
  - Intermountain Research Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - Wellborn Clinic, Evansville, Indiana
  - David Neustadt PSC, Louisville, Kentucky
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Great Lakes Research Group, Bay City, Michigan
  - Western Montana Clinic, Missoula, Montana
  - Physician Research Collaboration, Lincoln, Nebraska
  - Arthritis Center of Reno, Reno, Nevada
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Brian Gunnlaugson, MD, Johnstown, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, West Reading, Pennsylvania
  - SCRI, Germantown, Tennessee
  - Valley Orthopedic Clinic, Harlingen, Texas
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monovisc® | Saline
Started (Safety Population) | 184 | 185
Intend-to-treat ITT | 181 (3 of 184 excluded from ITT group for not having at least 1 post-injection visit. ITT=181 subjects) | 184 (1 of 185 excluded from ITT group for not having at least 1 post-injection visit. ITT=184 subjects)
Completed (Completed through 26 weeks follow-up) | 162 | 169
Not Completed | 22 | 16
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 7 | 6
Not completed — Use/Need of Con Therapy | 2 | 1
Not completed — Other - Reason Not Provided | 5 | 3

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Monovisc® | Saline | Total
Number analyzed (Participants) | 181 | 184 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (7.9) | 58.7 (9.2) | 59.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 106 | 213
  Male | 74 | 78 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 16 | 37
  White | 154 | 163 | 317
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score (ITT) >=40% and 15 mm From Baseline Through 12 Weeks
Description: The primary endpoint measures the percentage of subjects (Monovisc vs. saline) who achieved >= a 40% improvement (reduction) in the WOMAC Pain Score and show at least 15 mm improvement (reduction) in the WOMAC Pain Score from baseline through 12 weeks. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score is a validated scale from 0 to 100 mm, where a higher score is equal to a higher pain level. The primary endpoint uses the ITT population that has data available for both baseline and 12 week time points.
Time Frame: 12 Weeks
Population: Intent to Treat population includes all subjects who received a study injection and who had data for both baseline and 12 week time points.
Measure: Number; unit: Percentage of subjects
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 173 | 173
Percentage of subjects | 62.57 | 56.14
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.1450, Ordinal GEE Model

2. Secondary Outcome: Evaluator Global Assessment Change From Baseline Through Week 12 (ITT)
Description: Comparison of the change of the Evaluator Global Assessment from baseline through Week 12 between Monovisc and saline arms (ITT Population). The Evaluator Global Assessment is done by the Blinded Evaluator, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee affect him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a 0 to 100 mm Visual Analog Scale (VAS Scale), where a higher number means the patient is bothered to a higher degree. A negative number for the change from baseline indicates a reduction (improvement) in the assessment. The endpoint uses the ITT population that has data available for both baseline and 12 week time points.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 171 | 171
units on a scale
  Change from Baseline in Evaluator Global 12 weeks | -28.6 (26.4) | -26.4 (26.4)
  Baseline Evaluator Global | 59.1 (15.5) | 58.9 (14.6)
  12 Week Evaluator Global | 30.4 (23.5) | 32.1 (23.2)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.5824, Ordinal GEE Model

3. Secondary Outcome: Patient Global Assessment Change From Baseline Through Week 12 (ITT)
Description: Comparison of the change of the Patient Global Assessment from baseline through Week 12 between Monovisc and saline arms (ITT Population). The Patient Global Assessment is done by the patient, and answers the question "Considering all the ways the osteoarthritis in your study knee affects you, what is your assessment of how much your study knee is bothering you today?" The Patient Global Assessment is scored on a 0 to 100 mm Visual Analog Scale (VAS Scale), where a higher number means the patient is bothered to a higher degree. A negative number for the change from baseline indicates a reduction (improvement) in the assessment. The endpoint uses the ITT population that has data available for both baseline and 12 week time points.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 171 | 171
units on a scale
  Change from Baseline in Patient Global 12 weeks | -28.8 (30.8) | -28.9 (27.7)
  Baseline Patient Global | 62.9 (17.5) | 61.6 (16.7)
  12 Week Patient Global | 33.7 (25.0) | 33.2 (24.9)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.9136, Ordinal GEE Model

4. Secondary Outcome: Range of Motion Change From Baseline Through Week 12 (ITT)
Description: Comparison of the change of Range of Motion from baseline through Week 12 between Monovisc and saline arms (ITT Population). Range of motion is defined as the difference between flexion and extension in degrees where full extension range is 180 degrees. The endpoint uses the ITT population that has data available for both baseline and 12 week time points.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 171 | 171
degrees
  Change from Baseline in Range of Motion 12 weeks | 1.5 (14.9) | 4.6 (14.4)
  Baseline Range of Motion | 116.3 (16.4) | 114.5 (16.0)
  12 Week Range of Motion | 117.8 (14.4) | 119.3 (15.2)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.1699, Ordinal GEE Model

5. Secondary Outcome: WOMAC Physical Function Score Change From Baseline Through Week 12 (ITT)
Description: This endpoint compares the change of the WOMAC Physical Function Score from baseline through Week 12 between Monovisc and saline arms (ITT Population). The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Score is a validated scale from 0 to 100 mm, where a higher score is equal to a higher degree of functional limitation. A negative number for the change from baseline indicates improvement in physical function. The ITT population includes subjects with data at baseline and 12 Week time points.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 171 | 171
units on a scale
  Change from Baseline in WOMAC Function 12 weeks | -24.1 (26.1) | -22.3 (25.4)
  Baseline WOMAC Function | 55.8 (15.9) | 54.1 (17.3)
  12 Week WOMAC Function | 31.6 (26.2) | 31.7 (25.3)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.3238, Ordinal GEE Model

6. Post Hoc Outcome: Percentage Subjects Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score (ITT) >=50% and 20 mm From Baseline Through 26 Weeks
Description: This post-hoc endpoint measures the percentage of subjects (Monovisc vs. saline) who achieved >= a 50% improvement (reduction) in the WOMAC Pain Score and show at least 20 mm improvement (reduction) in the WOMAC Pain Score from baseline through 26 weeks. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score is a validated scale from 0 to 100 mm, where a higher score is equal to a higher pain level. Reduction in the WOMAC Pain Score from baseline (e.g. a negative number) indicates improvement in pain. The primary endpoint uses the ITT population that has data available for both baseline and 26 week timepoints.
Time Frame: 26 Weeks
Population: Intent-To-Treat population was defined as all randomized patients who received the study injection and had at least one post-injection visit; i.e: at least one visit after the Week 0 visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 171 | 171
Percentage of Participants | 44.38 | 34.12
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.0427, Ordinal GEE Model

7. Post Hoc Outcome: Evaluator Global Assessment Change From Baseline Through Week 26 (ITT)
Description: Comparison of the change of the Evaluator Global Assessment from baseline through Week 26 between Monovisc and saline arms (ITT Population). The Evaluator Global Assessment is done by the Blinded Evaluator, and answers the question "Considering all the ways the osteoarthritis in the patient's index knee affect him/her, what is your assessment of how much the patient's knee is bothering him/her today?" The Evaluator Global Assessment is scored on a 0 to 100 mm Visual Analog Scale, where a higher number means the patient is bothered to a higher degree. A negative number for the change from baseline indicates a reduction (improvement) in the assessment. The endpoint uses the ITT population that has data available for both baseline and 26 week time points.
Time Frame: 26 Weeks
Population: Intent to Treat population includes all subjects who received a study injection and who had data for both baseline and 26 week time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 162 | 168
units on a scale
  Change from Baseline in Evaluator Global 26 weeks | -27.9 (24.2) | -27.5 (27.5)
  Baseline Evaluator Global | 59.1 (15.5) | 58.9 (14.6)
  26 Week Evaluator Global | 31.9 (22.0) | 30.9 (22.9)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.8206, Ordinal GEE Model

8. Post Hoc Outcome: Patient Global Assessment Change From Baseline Through Week 26 (ITT)
Description: Comparison of the change of the Patient Global Assessment from baseline through Week 26 between Monovisc and saline arms (ITT Population). The Patient Global Assessment is done by the patient, and answers the question "Considering all the ways the osteoarthritis in your study knee affects you, what is your assessment of how much your study knee is bothering you today?" The Patient Global Assessment is scored on a 0 to 100 mm Visual analog Scale, where a higher number means the patient is bothered to a higher degree. A negative number for the change from baseline indicates a reduction (improvement) in the assessment. The endpoint uses the ITT population that has data available for both baseline and 26 week time points.
Time Frame: 26 Weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 162 | 168
units on a scale
  Change from Baseline in Patient Global 26 weeks | -28.5 (27.9) | -28.6 (27.2)
  Baseline Patient Global | 62.9 (17.5) | 61.6 (16.7)
  26 Week Patient Global | 33.7 (26.0) | 33.4 (26.2)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.9818, Ordinal GEE Model

9. Post Hoc Outcome: Range of Motion Change From Baseline Through Week 26 (ITT)
Description: Comparison of the change of Range of Motion from baseline through Week 26 between Monovisc and saline arms (ITT Population). Range of motion is defined as the difference between flexion and extension in degrees where full extension range is 180 degrees. The endpoint uses the ITT population that has data available for both baseline and 26 week time points.
Time Frame: 26 Weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 162 | 168
degrees
  Change from Baseline in Range of Motion 26 Weeks | 1.0 (14.9) | 4.2 (14.6)
  Baseline Range of Motion | 116.3 (16.4) | 114.5 (16.0)
  26 Week Range of Motion | 117.2 (13.9) | 118.8 (14.2)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.0542, Ordinal GEE Model

10. Post Hoc Outcome: WOMAC Physical Function Score Change From Baseline Through Week 26 (ITT)
Description: This endpoint compares the change of the WOMAC Physical Function Score from baseline through Week 26 between Monovisc and saline arms (ITT Population). The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Score is a validated scale from 0 to 100 mm, where a higher score is equal to a higher degree of functional limitation. A negative number for the change from baseline indicates improvement in physical function. The ITT population includes subjects with data at baseline and 26 Week time points.
Time Frame: 26 Weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monovisc® | Saline
Number analyzed (Participants) | 162 | 168
units on a scale
  Change from Baseline in WOMAC Function 26 weeks | -23.3 (26.0) | -21.4 (24.8)
  Baseline WOMAC Function | 55.8 (15.9) | 54.1 (17.3)
  26 Week WOMAC Function | 32.5 (24.8) | 33.1 (25.2)
Statistical Analysis 1: Comparison: Monovisc® vs Saline; Test type: Superiority; p = 0.3230, Ordinal GEE Model

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | Monovisc® | Saline
Serious Adverse Events (participants affected / at risk) | 9/184 | 5/185
Other Adverse Events (participants affected / at risk) | 121/184 | 123/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovisc® (N=184) | Saline (N=185)
Angina Unstable (Cardiac disorders) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovisc® (N=184) | Saline (N=185)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomach Discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (6) | 4 (7)
Influenza Like Illness (General disorders) | 2 (2) | 1 (1)
Injection Site Pain (General disorders) | 3 (3) | 1 (1)
Malaise (General disorders) | 1 (1) | 3 (3)
Oedema Peripheral (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 4 (5) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 5 (5) | 8 (8)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (9) | 11 (11)
Sinusitis (Infections and infestations) | 6 (7) | 5 (5)
Tooth Abscess (Infections and infestations) | 1 (1) | 2 (2)
Tooth Infection (Infections and infestations) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (14) | 14 (16)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 5 (6)
Back Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 6 (9) | 9 (11)
Excoriation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1) | 8 (8)
Muscle Strain (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (59) | 27 (44)
Back Pain (Musculoskeletal and connective tissue disorders) | 16 (26) | 16 (25)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9 (20) | 7 (7)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 15 (24) | 13 (14)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 24 (39) | 28 (56)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Migrane (Nervous system disorders) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 4 (4)
Sinus Headache (Nervous system disorders) | 4 (5) | 9 (14)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No